CLINICAL TRIAL: NCT06387706
Title: The Development of a Gamified Web-based Pain Management Program (GAP) for Community-dwelling Older Adults With Chronic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, TSE Mun Yee Mimi, Professor, Hong Kong Metropolitan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GAP
Record Dates: First submitted 2024-04-23; First posted 2024-04-29 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Chronic Pain Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GAP group (Experimental): Participants will be invited in the process of developing the GAP, the pain education materials, exercise videos, gameing elements and activities. Each stages of development of the GAP will be jointly monitored by the research team and the participants, feedback and comments will be constantly seek via biweekly meeting.
  Interventions: Other: Gamified web-based pain management Program

INTERVENTIONS:
Other: Gamified web-based pain management Program — Gamified Program Development: The project aims to create a Gamified web-based pain management Program (GAP) tailored for older adults with chronic pain, enhancing engagement through gaming elements.
  Inclusive Design Process: Older adults with chronic pain will actively participate in developing GAP, providing valuable feedback throughout the process.
  Pilot Study Design: A pre and post study design will be employed, with a small pilot group of 4 participants to offer diverse perspectives in the program's development.
  Educational Content & Activities: GAP will feature interactive educational content on pain effects, medication, non-drug treatments, and exercises, delivered through a mobile-friendly web platform.

SUMMARY:
Pain Management in Older Adults: Pain significantly impacts the well-being of older adults, often leading to diminished physical abilities and a reduced quality of life. Despite this, pain management remains suboptimal, with concerns about medication side effects and a tendency to view pain as a natural aspect of aging. Consequently, many seniors are hesitant to use painkillers. As an alternative, non-pharmacological strategies such as educational programs, physical activity, massage, relaxation techniques, and music therapy are gaining traction.

Innovative Non-Drug Solutions: To improve participation in non-medication pain relief methods, we suggest incorporating gaming elements into these programs (GAP). Originating in digital media in 2008, gamification has since spread across various industries. It involves adding game-like elements to activities to boost engagement, experience, and motivation.

Project Goals: The aims of this initiative include creating a web-based Gamified Pain Management Program (GAP), engaging older adults with chronic pain in the development of GAP, and gathering their feedback on the program's effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 or above
* Can understand Cantonese
* Scored >6 in the Abbreviated Mental Test; a cut-off point of 6 is valid for differentiating between normal and abnormal cognitive functions in geriatric clients
* Have a history of non-cancer pain in the past 6 months
* Have a pain score of at least 2 on the Numeric Rating Scale
* Able to take part in light exercise and stretching
* Owns a smartphone and can access the Internet

Exclusion Criteria:

* Have severe visual and/or auditory deficits that affect that seeing and hearing
* Have a serious organic disease or malignant tumor
* Have a mental disorder diagnosed by neurologists or psychiatrists
* Had a surgical treatment in the past two months
* Experienced drug addiction

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Pain Relief | 4-week
  Conducting pre- and post-test of Brief Pain Inventory Scale Title: Brief Pain Inventory Minimum Value: 0 Maximum Value: 10 Interpretation: Higher scores indicate worse pain outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Metropolitan University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No